CLINICAL TRIAL: NCT02029105
Title: PREDICTING MALIGNANT MESOTHELIOMA BY ANALYZING HYALURONAN, OSTEOPONTIN, C-ERC/MESOTHELIN, N-ERC/MESOTHELIN AND SYNDECAN-1 SERUM LEVELS
Brief Title: Serum Biomarkers in Diagnosis of Mesothelioma
Status: Completed | Type: Observational
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Muzaffer Metintas, Eskisehir Osmangazi University Lung and Pleural Cancers Application and Research Center-Turkey; Director, Eskisehir Osmangazi University
Other Study IDs: 2010-280-1
Record Dates: First submitted 2014-01-06; First posted 2014-01-07 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: Mesothelioma
Keywords: Mesothelioma,; Pleural diseases,; Mesothelin,; Osteopontin,; Hyaluronan,; Syndecan-1
MeSH Terms: conditions — Mesothelioma; Pleural Diseases | interventions — Mesothelin; Hyaluronic Acid; Osteopontin; Syndecan-1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Serum samples of the patients
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Mesothelin, hyaluronan, osteopontin, syndecan: The patients with pleural diseases
  Interventions: Biological: Mesothelin, hyaluronan, osteopontin, syndecan-1

INTERVENTIONS:
Biological: Mesothelin, hyaluronan, osteopontin, syndecan-1 — We compere the serum levels of the tumor markers in patients with pleural diseases according to the groups for the diagnosis and differential diagnosis of the diseases.
  Other Names: N-ERC/mesotehlin,; C-ERC/mesotehlin; Osteopontin; Hyaluronan; Syndecan-1

SUMMARY:
In this study, the investigators analyzed the efficiencies of hyaluronan, osteopontin, C-ERC/mesothelin, N-ERC/mesothelin and syndecan-1 serum levels, both individually and in combination, in distinguishing malignant pleural mesothelioma patients from patients with metastatic malignant pleural diseases, benign pleural diseases, and benign asbestos pleurisy.

DETAILED DESCRIPTION:
In the year 2002, a database for the pleural diseases was constructed to be prospectively filled in the department. The findings, outcome features and characteristics of follow-up for all cases with pleural diseases have been recorded in this database. The patient data, including epidemiological characteristics, smoking status, history of other diseases and co-morbid conditions, previous asbestos exposure, medications and additional physical and radiological examination findings, including computed tomography scans, both serum and pleural fluid laboratory investigational data and indications of invasive procedures, were recorded in the database mentioned above. The methods employed in the diagnosis of patients; any complications; characteristics such as the stages of diseases, treatments, and course of treatments; and results were also recorded in the database. From the date of the first database establishment, a "tissue, blood, serum, and fluid specimen bank" was constructed; tissue, blood, serum and pleural fluid samples of patients, which had been taken at the beginning of diagnosis process, were stored in this bank at -80°C. The blood, serum, and pleural fluid samples of patients were stored during the diagnosis process, and if conducted, pleural tissue samples taken during invasive procedures were also stocked.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a definite pleural diseases
* Age more than 18 year-old, less than 85 year-old.
* Willingness to participate in the study.

Exclusion Criteria:

* Patients with undiagnosed pleural diseases.
* Age less than 18 year-old or more than 85 year-old.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pleural diseases; mesothelioma, metastatic malignant pleural diseases, benign pleural diseases and benign asbestos pleurisy.
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2004-01; Primary Completion 2010-12 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Serum N-ERC/mesothelin, C-ERC/mesothelin, hyaluronan, osteopontin and syndecan -1 level in the patients with mesothelioma, metastatic malignant pleural diseases, benign pleural diseases, and benign asbestos pleurisy. | From January 2004 to December 2010
  The levels of N-ERC/mesothelin, C-ERC/mesothelin, hyaluronan, osteopontin, and syndecan-1 in the serum samples were established by Enzyme-Linked Immunosorbent Assays (ELISA) at the Division of Pathology, Department of LABMED, Karolinska Institute, Stockholm, Sweden.
  All analyses were performed in duplicate by researchers who were unaware of the patient diagnoses. The human N-ERC/mesothelin and osteopontin. ELISA kits were supplied by Immuno-Biological Laboratories Co. Ltd. Japan; the C-ERC/mesothelin ELISA kit was supplied by (MESOMARK™) FDI Fujirebio Diagnostics, Inc.; the hyaluronan ELISA kit (Ref. 029-001) was supplied by Corgenix company; and the syndecan-1 ELISA kit (catalog no. 950.640.096) was supplied by the Diaclone company. Analyses were conducted using a sensitivity TM XS Microplate Sample Processor manufactured by Bio-Tek Instruments Inc (Vermont, USA) in accordance with the manufacturer's instructions. The C-ERC/mesothelin levels were determined at nanomolar levels due

CONTACTS AND LOCATIONS:
Overall Officials: Muzaffer Metintas, Prof.Dr., Study Director — Eskisehir Osmangazi University
Locations (1):
- ESOGU Lung and Pleural Cancer Application and Research Center, Eskişehir, Turkey (Türkiye)